CLINICAL TRIAL: NCT02046538
Title: Phase II Study of Preoperative Chemotherapy With Ziv-aflibercept (Zaltrap) Followed by Postoperative Chemotherapy With or Without Ziv-aflibercept (Zaltrap) in Patients With Advanced Resectable Colorectal Cancer
Brief Title: Phase II Study of Zaltrap and Chemotherapy for Advanced Resectable Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator terminated due to funding issues
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1309014302; 2012-AFL-18 (Other Grant/Funding Number: Sanofi)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Leucovorin; Oxaliplatin; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postoperative Chemo WITH Zaltrap (Experimental): Subjects will receive 3 months of chemotherapy consisting of either FOLFOX (oxaliplatin, leucovorin, 5-FU) or FOLFIRI (Irinotecan, leucovorin, 5-FU) in the case of liver limited CRC, or FOLFOX (in the case of rectal cancer). Zaltrap will be administered with chemotherapy every 2 weeks for the first 5 out of 6 planned treatment cycles. After a standard 3-4 week recovery period (i.e. 5-6 weeks from the last Zaltrap dose), patients will undergo standard resection. At the time of resection, the tumor will be collected for biomarker discovery.
  Following resection, patients will receive chemotherapy with zaltrap for 3 additional months. Patients may continue zaltrap (without chemotherapy) until disease recurrence or up to an additional 15 months.
  Interventions: Drug: Leucovorin; Drug: Oxaliplatin; Drug: 5-FU; Drug: Irinotecan
- Postoperative chemo WITHOUT zaltrap (Active Comparator): Subjects will receive 3 months of chemotherapy consisting of either FOLFOX (oxaliplatin, leucovorin, 5-FU) or FOLFIRI (Irinotecan, leucovorin, 5-FU) in the case of liver limited CRC, or FOLFOX (in the case of rectal cancer). Zaltrap will be administered with chemotherapy every 2 weeks for the first 5 out of 6 planned treatment cycles. After a standard 3-4 week recovery period (i.e. 5-6 weeks from the last Zaltrap dose), patients will undergo standard resection. At the time of resection, the tumor will be collected for biomarker discovery.
  Following resection, patients will receive chemotherapy (without zaltrap) for 3 additional months.
  Interventions: Drug: Leucovorin; Drug: Oxaliplatin; Drug: 5-FU; Drug: Irinotecan

INTERVENTIONS:
Drug: Leucovorin — 400 mg/m2 IV over two hours (or administered concurrently with oxaliplatin or irinotecan, depending on the assigned regimen)
  Other Names: Wellcovorin
Drug: Oxaliplatin — 85 mg/m2 IV over two hours
  Other Names: Eloxatin
Drug: 5-FU — 400 mg/m2 IV bolus, then 2400 mg/m2 continuous IV infusion over 46-48 hours
  Other Names: Adrucil, fluorouracil
Drug: Irinotecan — 180 mg/m2 IV over 90 minutes
  Other Names: Camptosar

SUMMARY:
The purpose of this study is to establish the safety of Zaltrap in patients who undergo pre-operative chemotherapy with Zaltrap. The investigators hypothesize that Zaltrap my impact colorectal cancer growth and metastasis.

DETAILED DESCRIPTION:
Eligible patients will receive 3 months of chemotherapy consisting of either FOLFOX or FOLFIRI (in the case of liver limited CRC) or FOLFOX (in the case of rectal cancer). The FOLFOX regimen consists of Oxaliplatin, Leucovorin, and 5-FU. The FOLFIRI regimen consists of Irinotecan, Leucovorin, and 5-FU. Zaltrap will be administered with chemotherapy every 2 weeks for the first 5 out of 6 planned treatment cycles. After a standard 3-4 week recovery period (i.e. 5-6 week's from the last Zaltrap dose), patients will undergo standard resection. At the time of resection, the tumor will be collected for biomarker discovery.

Following resection, patients will be randomly assigned (1:1) to receive chemotherapy with or without zaltrap for 3 additional months. Patients assigned to Zaltrap may continue zaltrap (without chemotherapy) until disease recurrence or up to an additional 15 months. Patients will have research blood draws periodically both in the preoperative and postoperative period.

The investigators plan to demonstrate that pre-operative chemotherapy with Zaltrap is not associated with any safety signals that would preclude further drug development in this patient population. The investigators also plan to perform correlative studies to identify potential biomarkers for Zaltrap activity.

The investigators hypothesize that antiangiogenic therapy may specifically target the micrometastatis niche of patients with liver limited metastatic colorectal cancer to significantly increase the chance of cure for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed adenocarcinoma of the colon or rectum.
* In patients with liver-limited metastatic colorectal cancer, a curative approach is indicated following evaluation by hepatobiliary surgeon as part of multidisciplinary management. Select patients requiring two stage procedure are also eligible following evaluation by hepatobiliary surgeon as part of multidisciplinary management.
* In patients with rectal cancer, primary tumor that is clinically T3-4 or N + (evaluation by colorectal surgery is required as part of multidisciplinary approach).
* No prior chemotherapy for metastatic disease is allowed for patients with CRC-liver mets. (adjuvant FOLFOX is permitted)
* No prior chemotherapy for proximal rectal cancer is allowed
* ECOG Performance status ≤ 2.
* Age >18 years old.
* Patients must have adequate bone marrow, kidney, and liver function as assessed by laboratory parameters.

  1. WBC ≥ 3,000/uL
  2. Total Bilirubin ≤ 1.5 x upper limits of normal
  3. AST (SGOT) ≤ 3 x upper limits of normal
  4. ALT (SGPT) ≤ 3 x upper limits of normal
  5. Hemoglobin ≥ 9.0 g/dl (without transfusion within 7 d)
  6. ANC ≥ 1500 /ml
  7. Platelets ≥100 K/ml (without transfusion)
  8. Calculated CrCL > 50 ml/min
* Ability to understand and the willingness to sign a written informed consent document.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Patients with untreated CNS metastases.
* Significant medical co-morbidity that would preclude safe administration of cytotoxic therapy, including but not limited to:

  1. Cardiovascular disease

     1. Unstable angina
     2. Myocardial infarction/ CABG < 3 months prior to study initiation
     3. Untreated coronary artery disease
     4. NYHA class III or IV heart failure
  2. Ongoing serious infection

     1. Bacteremia or sepsis requiring intravenous antibiotics
     2. HIV with AIDS defining illness
  3. Inadequate oral nutritional intake: Requirement for daily intravenous fluids or total parenteral nutrition.
  4. Neurological: Stroke ≤ 6 months
  5. Psychiatric illness/social situations that would limit compliance with study requirement
* Patients may not receive another investigational agent.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Ziv-aflibercept.
* Pregnant (positive pregnancy test) and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.
* Major surgical procedure ≤ 4 weeks from starting therapy.
* Grade 3-4 hemorrhage, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulits ≤ 3 months from starting therapy.
* Patients with known DPD deficiency
* Patients with known Gilbert's syndrome
* Patients with ≥ 2g/24 hour urine protein. If urine protein on random UA is ≤ 300 mg/dl, a 24 hour urine protein is not required.
* Symptomatic peripheral sensory neuropathy grade ≥ 2.
* Other malignancy within the last 5 years from study entry, except for basal /squamous cell skin cancer, in situ cervical cancer, or non-metastatic prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events experienced | Approximately 24 months per patient
  Capture the number of adverse events experienced by advanced resectable colorectal cancer subjects treated with pre-operative chemotherapy and Zaltrap
Number of subjects who demonstrate a response to pre-operative chemotherapy and zaltrap | Approximately 24 months per patient
  Capture the number of subjects who demonstrate an improvement (response) in colorectal cancer status after being treated with pre-operative chemotherapy and zaltrap.

SECONDARY OUTCOMES:
Survival duration without disease progression | 2 years per patient
  Calculate rate of progression-free survival for subjects following treatment chemotherapy and Zaltrap

CONTACTS AND LOCATIONS:
Overall Officials: Manish A. Shah, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No